CLINICAL TRIAL: NCT01174576
Title: Acute Effects of Caffeinated and Decaffeinated Coffee Consumption on Energy Intake, Appetite, Inflammation and Glucose Metabolism
Brief Title: Acute Effects of Coffee on Appetite and Inflammation Markers, Glucose Metabolism and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, M. Yannakoulia, PhD, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CofSt
Record Dates: First submitted 2010-07-26; First posted 2010-08-03 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-07

CONDITIONS: Health
Keywords: coffee; appetite; energy intake; inflammation; cortisol; glucose; randomized controlled trial
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- caffeinated coffee (Experimental): 200 mL caffeinated coffee with 3 mg caffeine per kg body weight
  Interventions: Other: caffeinated and decaffeinated coffee
- decaffeinated coffee (Experimental): 200 mL decaffeinated coffee, same amount as caffeinated coffee
  Interventions: Other: caffeinated and decaffeinated coffee
- Water (Experimental): 200 mL, control intervention
  Interventions: Other: caffeinated and decaffeinated coffee

INTERVENTIONS:
Other: caffeinated and decaffeinated coffee — 3 treatments on separate days, i.e. a standard breakfast with oral ingestion of 200 ml of either caffeinated coffee (3mg caffeine/kg body weight), decaffeinated coffee or water

SUMMARY:
The purpose of the study is to investigate whether caffeinated and decaffeinated coffee consumption has acute effects on subjective appetite feelings, energy intake and biochemical markers related to appetite, inflammation and glucose metabolism compared to water consumption.

DETAILED DESCRIPTION:
Coffee is a pharmacologically active, widely consumed beverage. Scientific interest in relation to coffee consumption has been revisited the last decade in the light of new, mainly epidemiological, evidence indicating its potential health benefits. In specific, both cross-sectional and prospective studies indicate that coffee consumption is associated with a lower risk for type 2 diabetes. Furthermore, an inverse association has been found between coffee consumption and markers of inflammation and endothelial dysfunction in healthy and/or diabetic participants, although the opposite effect has also been reported, mainly in relation to inflammation markers. In relation to body weight, epidemiological data suggest that increment in caffeine consumption is associated with lower mean weight gain and energy intake during a 12-y period.

However, information from clinical studies is scarce. Acute caffeine and/or coffee consumption have been associated with impaired glucose metabolism and insulin resistance. In relation to inflammation, animal studies have indicated a beneficial or no effect of coffee consumption, whereas a clinical study in humans found an increase in adiponectin and a decrease in interleukin-18 (IL-18) blood concentrations after a monthly intervention including daily consumption of 8 cups of coffee. As far as energy balance is concerned, there is an early experiment demonstrating that the ingestion of 300 mg of caffeine prior to food intake, compared to the non-caffeine intake, significantly reduced energy intake by 21.7% in men, but not in women. A more recent study has found that the combination of caffeine and red pepper is positively associated with energy expenditure and negatively with energy intake, whereas, it has also been reported a positive association between habitual caffeine intake and body weight loss achieved through a very-low-calorie diet.

Taking into consideration the limited clinical evidence regarding the acute effect of coffee consumption on appetite-related markers, subsequent energy intake and inflammatory markers, we undertook a clinical study of crossover design to investigate the short-term changes on energy intake, subjective appetite ratings, appetite hormones, inflammation markers and glucose metabolism after caffeinated and decaffeinated coffee consumption.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-obese

Exclusion Criteria:

* smokers
* restrained eaters (as this was evaluated using the Dutch Eating Behaviour Questionnaire and a total score > 2.5)
* those who reported slimming or any other dietary regime
* abstainers from caffeine sources
* athletes during competition period
* participants with a known diagnosis of either hypertension, diabetes, impaired glucose tolerance or a fasting blood glucose concentration above 125 mg/dl
* subjects on medication for hypertension or on medication known to alter glucose metabolism
* subjects who were on medication that may have an impact on appetite and sensory functioning or who reported a metabolic or endocrine disease, gastrointestinal disorders, or a history of medical or surgical events that may have affected the study outcomes

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Yannakoulia, PhD, Study Director — Harokopio University
Locations (1):
- Metabolic Unit of the Department of Nutrition and Dietetics, Harokopio University, Athens, Greece

REFERENCES:
- [Derived] Gavrieli A, Yannakoulia M, Fragopoulou E, Margaritopoulos D, Chamberland JP, Kaisari P, Kavouras SA, Mantzoros CS. Caffeinated coffee does not acutely affect energy intake, appetite, or inflammation but prevents serum cortisol concentrations from falling in healthy men. J Nutr. 2011 Apr 1;141(4):703-7. doi: 10.3945/jn.110.137323. Epub 2011 Feb 23. PMID 21346100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February-Mai 2009, Athens region, voluntarily recruitment
Groups:
- Caffeinated Coffee/Decaffeinated Coffee/Water: 200 ml instant caffeinated coffee with 3 mg caffeine/kg body weight or instant decaffeinated coffee or water. All participants received all interventions without exception in a random order.
  Three combinations of treatment sequences were used:
  1. Caffeinated coffee, then decaffeinated coffee, then water
  2. Decaffeinated coffee first, then water, then caffeinated coffee
  3. Water first, then caffeinated coffee, then decaffeinated coffee.
  Each treatment was separated by the other by at least one week interval.
  The first volunteer entered the study received the first combination, the second volunteer the second combiation, the third volunteer the third combination, the forth volunteer the first combination of treatments, etc.
Period: Overall Study
Arm/Group | Caffeinated Coffee/Decaffeinated Coffee/Water
Started | 16 (All participants received all interventions without exception.)
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Region of Enrollment [Number; unit: participants]
  Greece | 16

OUTCOME MEASURES:

1. Primary Outcome: Ghrelin Total Area Under the Curve
Description: Total area under the curve was defined as the sum of the areas under and over the baseline using the trapezoidal rule. The time points for the calculations were 15 min before beverage consumption, immediately after beverage consumption, 15, 30, 60, 90, 120, 150, 180 min postconsumption.
Time Frame: 15 min before ingestion to 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: ug*h/mL
Groups:
- Caffeinated Coffee: 200 mL, 3 mg caffeine/kg body weight
- Decaffeinated Coffee: 200 mL, same amount as caffeinated coffee
- Water: 200 mL
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
ug*h/mL | 2669 (786) | 2593 (778) | 2672 (902)

2. Primary Outcome: Peptide Tyrosine Tyrosine (PYY) Total Area Under the Curve
Description: as for outcome 1
Time Frame: 15 min before ingestion to 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
pg*h/mL | 251 (136) | 286 (138) | 259 (158)

3. Primary Outcome: Glucagon-like Peptide-1 (GLP-1) Total Area Under the Curve
Description: as for outcome 1
Time Frame: 15 min before ingestion to 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
ug*h/mL | 43 (61) | 45 (69) | 61 (122)

4. Primary Outcome: Adiponectin Total Area Under the Curve
Description: as for outcome 1
Time Frame: 15 min before ingestion to 3 h post ingestion
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
ug*h/mL | 22.7 (8.8) | 22.6 (10.2) | 22.6 (11.0)

5. Primary Outcome: Inteleukin-6 Total Area Under the Curve
Description: as for outcome 1
Time Frame: 15 min before ingestion to 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: pg*h/mL
Groups:
- Decaffeinated Coffee: 200 mL, same amount as caffeineated coffee
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
pg*h/mL | 5.4 (2.1) | 5.5 (2.5) | 6.0 (2.6)

6. Primary Outcome: Interleukin-18 Total Area Under the Curve
Description: as for outcome 1
Time Frame: 15 min before ingestion to 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
pg*h/mL | 818 (289) | 777 (280) | 786 (273)

7. Primary Outcome: Glucose Total Area Under the Curve
Description: as for outcome 1
Time Frame: 15 min before ingestion to 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: mg*h/dl
Groups:
- Caffeinated Coffee: 200 ml instant caffeinated coffee with 3 mg caffeine/kg body weight
- Decaffeinated Coffee: 200 ml instant decaffeinated coffee
- Water: 200 ml water
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
mg*h/dl | 336 (22) | 329 (20) | 323 (20)

8. Secondary Outcome: Serum Antioxidant Capacity Total Area Under the Curve
Description: Serum samples, collected 15 min before ingestion, immediately after ingestion, 15 min, 30 min, 60 min, 90 min, 120 min and 150 min after ingestion were analyzed for the ex vivo serum resistance to oxidative stress, that was induced by copper sulfate (CuSO4). The analysis of all collected samples was performed by the measurement of conjugated diene formation, which was monitored for every sample of all time points every 2 min for a 3.5 h period at 234 nm in a microplate spectrophotometer.
  Total area under the curve was defined as the sum of the areas under and over the baseline using the trapezoidal rule. The time points for the calculations were 15 min before beverage consumption, immediately after beverage consumption, 15, 30, 60, 90, 120, 150 min postconsumption.
Time Frame: 15 min before ingestion to 21/2 hr post ingestion
Measure: Mean (Standard Deviation); unit: lag time (min) *h
Groups:
- Caffeinated Coffee: 200 mL, 3 mg caffeine/ kg body weight
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
lag time (min) *h | 102 (30) | 104 (37) | 108 (32)

9. Primary Outcome: Insulin Total Area Under the Curve
Description: as for outcome 1
Time Frame: 15 min before ingestion to 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: uU*h/ml
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
uU*h/ml | 54 (14) | 52 (16) | 52 (16)

10. Primary Outcome: Cortisol Total Area Under the Curve
Description: as for outcome 1
Time Frame: 15 min before ingestion to 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: ug*h/dL
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
ug*h/dL | 43.2 (11.3) | 39.8 (10.5) | 35.0 (6.9)

11. Primary Outcome: Energy ad Libitum Meal
Description: The energy of first meal 3 hr after ingestion
Time Frame: 3 hr post ingestion
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
kcal | 1749 (407) | 1720 (402) | 1750 (442)

12. Primary Outcome: Total Energy Intake
Description: the energy consumed at breakfast, ad libitum meal and rest of the experimental day
Time Frame: 1 d
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Number analyzed (Participants) | 16 | 16 | 16
kcal | 3223 (735) | 3445 (871) | 3302 (971)

ADVERSE EVENTS:
Time Frame: 3 h
Description: blood pressure and heart rate assessment
Groups:
- Caffeinated Coffee: 200 mL, coffee containing 3 mg caffeine/kg body weight
Arm/Group | Caffeinated Coffee | Decaffeinated Coffee | Water
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
the results cannot be generalized to other population groups, as participants were selected according to specific criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No